CLINICAL TRIAL: NCT03568929
Title: Non-interventional Study to Assess the Safety Profile of Idelalisib in Patients With Refractory Follicular Lymphoma (FL)
Brief Title: Safety Profile of Idelalisib in Patients With Refractory Follicular Lymphoma
Acronym: ZEUS
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-EU-313-4172; EUPAS19618 (Other: ENCePP)
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Follicular Non-Hodgkin's Lymphoma Refractory
MeSH Terms: interventions — idelalisib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Idelalisib: Participants who have been or are currently being treated with 100 or 150 mg of idelalisib
  Interventions: Drug: Idelalisib

INTERVENTIONS:
Drug: Idelalisib — Tablets administered according to the product information and treatment guidelines in routine clinical practice
  Other Names: Zydelig®

SUMMARY:
The primary objective of this study is to assess the overall safety profile of idelalisib monotherapy in patients with refractory follicular lymphoma (FL).

ELIGIBILITY:
Inclusion Criteria:

* Individuals who were or are being treated for refractory Follicular Lymphoma (FL) according to the product information for idelalisib and treatment guidelines in routine clinical practice.

Exclusion Criteria:

* Individuals included in clinical trials on idelalisib within the timeframe of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who were or are being treated with idelalisib for refractory FL according to the product information and treatment guidelines in routine clinical practice after the country specific approval date.
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Overall Safety Profile of Idelalisib as Measured by the Incidence of Adverse Events (AE), Serious AEs, Special Situation Reports, Adverse Drug Reactions (ADR), and Serious ADRs | 250 patient-years (8 months of treatment period, 3 years of retrospective time frame, and 2.5 years of prospective observation period)

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 250 patient-years (8 months of treatment period, 3 years of retrospective time frame, and 2.5 years of prospective observation period)
  ORR is defined as the proportion of participants who achieve a clinical response with or without radiological confirmation as documented within their electronic health record after the initiation of treatment with idelalisib and during the treatment period with idelalisib.
Duration of Response (DOR) | 250 patient-years (8 months of treatment period, 3 years of retrospective time frame, and 2.5 years of prospective observation period)
  DOR is defined as the interval from the first documentation of a clinical response with or without radiological confirmation to the earlier of the first documentation of disease progression or death from any cause.
Progression-free Survival (PFS) | 250 patient-years (8 months of treatment period, 3 years of retrospective time frame, and 2.5 years of prospective observation period)
  PFS is defined as the interval from the date of initiation of idelalisib to the earlier date of the first documentation of disease progression or death from any cause.
Time to Next Treatment (TTNT) | 250 patient-years (8 months of treatment period, 3 years of retrospective time frame, and 2.5 years of prospective observation period)
  TTNT is defined as the interval from the initiation of treatment with idelalisib to the earlier date of the initiation of next systemic treatment of Follicular Lymphoma (excluding palliative care or palliative radiation) or death from any cause.
Overall Survival (OS) | 250 patient-years (8 months of treatment period, 3 years of retrospective time frame, and 2.5 years of prospective observation period)
  OS is defined as the interval from the date of initiation of idelalisib to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (88):
- Ziekenhuis Netwerk Antwerpen Stuivenberg Hospital, Antwerp, Belgium
- France (17):
  - Centre Hospitalier Universitaire d'Amiens (CHU d'Amiens) - Hopital Nord, Amiens
  - Centre Hospitalier Bourg-en-Bresse Fleyriat, Bourg-en-Bresse
  - Centre Hospitalier de Cannes, Cannes
  - Hôpital Privé Sévigné, Cesson-Sévigné
  - Centre Hospitalier Chalon sur Saône William Morey, Chalon-sur-Saône
  - Centre Hospitalier Universitaire Estaing, Clermont-Ferrand
  - CHU de Dijon, Dijon
  - Groupe Hospitalier Mutualiste de Grenoble - Institut Daniel Hollard, Grenoble
  - Clinique Victor Hugo, Le Mans
  - Centre Hospitalier Le Mans, Le Mans
  - Centre Hospitalier de Lens, Lens
  - Hôpital de la Conception, Marseille
  - Centre Hospitalier Régional d'Orléans, Orléans
  - Centre hospitalier de Perigueux, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Hopital Bretonneau, Centre Henri Kaplan, Tours
- Germany (4):
  - Klinikum Frankfurt Hochst, Frankfurt
  - Universitätsmedizin Göttingen, Göttingen
  - Klinikum Südstadt Rostock, Rostock
  - Gemeinschaftspraxis für Hämatologie und Onkologie Westerstede, Westerstede
- Greece (5):
  - University General Hospital of Alexandroupolis, Alexandroupoli
  - Athens Medical Center-Psychikon branch, Athens
  - Henry Dunant Hospital, Athens
  - University General Hospital of Patras, Pátrai
  - AHEPA University General Hospital of Thessaloniki, Thessaloniki
- Ireland (3):
  - Saint James's Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - Midland Regional Hospital - Mullingar, Mullingar
- Italy (27):
  - Ospedali Riuniti di Ancona, Clinica Ematologica, Ancona
  - Ospedale Mazzoni, Ascoli Piceno
  - Azienda Ospedaliera Policlinico di Bari, Bari
  - Monsignor Raffaele Dimiccoli Hospital, Barletta
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera di Rilievo Nazionale e di Alta Specializzazione Garibaldi, Catania
  - Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele, Catania
  - Ospedale di Civitanova Marche, Civitanova Marche
  - Azienda Ospedaliero - Universitaria Careggi, Florence
  - Presidio Ospedaliero di Livorno, Livorno
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Fondazione IRCCS Cà Grande Ospedale Maggiore Policlinico, Milan
  - Istituto Scientifico Universitario San Raffaele, Milan
  - Azienda Ospedaliera Universitaria Maggiore Della Carita di Novara, Novara
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera di Perugia, Perugia
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Pesaro
  - Azienda Unità Sanitaria Locale di Piacenza-Ospedale Guglielmo da Saliceto, Piacenza
  - Azienda Unita Sanitaria Locale di Ravenna, Ravenna
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - IRCCS Centro di Riferimento Oncologico di Basilicata di Rionero in Vulture, Rionero in Vulture
  - Universita degli Studi di Roma La Sapienza, Roma
  - Istituti di Ricovero e Cura A Carattere Scientifico - Istituti Fisioterapici Ospitalieri, Roma
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Azienda Ospedaliera Universitaria Senese-L'ospedale Santa Maria alle Scotte, Siena
  - Ospedale San Bortolo di Vicenza, Vicenza
- Instituto Português de Oncologia Francisco Gentil, Centro Regional de Lisboa SA, Lisbon, Portugal
- Spain (25):
  - Fundació Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Universitari Mútua Terrassa, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital De Cabuenes, Gijón
  - Hospital Universitario Donostia, Gipuzkoa
  - Institut Català d'Oncologia, L'Hospitalet de Llobregat
  - Hospital Universitario Severo Ochoa, Leganés
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital San Pedro de Alcantara, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Rey Juan Carlos, Móstoles
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Son Dureta, Palma de Mallorca
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitari Arnau De Vilanova (Huav), Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
  - Hospital de Día Quirónsalud Zaragoza, Zaragoza
- Karolinska Universitetssjukhuset, Stockholm, Sweden
- United Kingdom (4):
  - Velindre NHS Trust, Cardiff
  - St George's Healthcare NHS Trust, London
  - South Tees Hospitals Nhs Foundation Trust, Middlesbrough
  - Abertawe Bro Morgannwg University Health Board, Swansea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-EU-313-4172